CLINICAL TRIAL: NCT01846767
Title: Study of the Metabolism of 13C Labelled Glucose to 13CO2 in Human Breath
Brief Title: Exogenous Glucose Oxidation Breath Test
Acronym: EGOBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Irish Endocrine Society (Other)
Responsible Party: Principal Investigator, Amir Shafat, Dr, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 13CGLU
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: 13CO2; Breath test; Glucose oxidation; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Type 2 diabetes (Experimental): Diabetic patients Oral glucose breath test
  Interventions: Other: Oral glucose breath test
- Healthy controls (Experimental): non-diabetic Oral glucose breath test
  Interventions: Other: Oral glucose breath test

INTERVENTIONS:
Other: Oral glucose breath test — Simultaneous oral glucose tolerance test and exogenous 13C-glucose breath test following a 12hr overnight fast. Fasting samples were obtained for plasma glucose, insulin, c-peptide, leptin, adiponectin, resistin, HbA1c and two breath 13CO2 abundance values (at t = -15 and -5min). At t = 0min, each subject drank a 75g glucose solution (Thornton & Ross, UK) containing 0.15g of 1-13C glucose. Further breath samples (every 15 min over a 240min interval) and further plasma blood glucose, insulin and c-peptide samples (90,120,180min) were also taken.

SUMMARY:
The purpose of this study is to determine if oxidation of 13C glucose to 13CO2 is changed in type 2 diabetic patients.

DETAILED DESCRIPTION:
Recruitment

- Non diabetic participants will be recruited from within the National University of Ireland, Galway student and staff community. Diabetic patients will be recruited from University College Hospital, Galway in collaboration with their hospital consultant.

Test- day

- They will undergo two separate, identical and simultaneous Oral Glucose Tolerance test and 13C-glucose breath tests on two separate occasions after an overnight fast of 12 hours starting at 8pm. On arrival their heart rate, blood pressure, height and weight will be recorded. Following a resting period of 10 minutes, samples will be obtained for fasting glucose and breath enrichment values (at t = -20 and -10mins). At t = 0 min, participants will consume a standard glucose solution. This glucose solution will consist of 150mg of 13C-glucose, 74.85g of glucose and 200ml of water and 25ml of orange flavoring. Breath samples will be obtained immediately after consumption of test solution and repeated every 15 min over a 4-h interval. Blood glucose concentrations will be taken every 15 min starting at t = 15 min, over a 2-h interval and every 30 min for another 2-h interval. Participants will remain at rest throughout the study.

Sample size assessment

- Target recruitment is 40 non-diabetics and 40 diabetic participants. This study will use a Student's t-test to determine difference, or otherwise, in glucose oxidation in breath 13CO2, in 2 different groups of individuals. With power arbitrarily set at 0.8, effect size of 1.21 reduction in breath, and Alpha set at 0.01 a final number of 35 participants is required for each group. The n=40 for each group is set to allow a 5 participant drop out in each group Dillon et al (2009).

ELIGIBILITY:
Inclusion Criteria:

* All research participants must be between 18 and 65 years
* Non-diabetic participants must not be taking any medication for diabetes
* Participants must speak English or Irish proficiently
* All participants must be males
* All participants must live within Galway City
* Type 2 diabetic participants must have been diagnosed within the last five years
* Type 2 diabetic participants must be treated by Metformin alone for their diabetes
* All participants must provide written informed consent to comply with every aspect of the study

Exclusion Criteria:

* Females

Ages: 35 Years to 82 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Peak Delta over baseline in 13CO2 breath enrichment | at 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240 minutes after glucose ingestion.
  The peak enrichment of 13CO2 in breath is calculated by identifying the highest abundance breath sample and subtracting the base line abundance from it.

SECONDARY OUTCOMES:
Per cent dose recovered | 240 minutes
  The per cent dose recovered of 13C glucose at 240 minutes.

OTHER OUTCOMES:
Diabetes classifications and measures of insulin resistance | 0 and 120 minutes
  Fasting plasma glucose and glucose tolerance at 120min, as defined by plasma glucose concentrations. Also measured Leptin/Adiponectin concentrations, Fasting insulin, calculated homeostatic model assessment and and quantitative insulin sensitivity check index.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Shafat, PhD, Principal Investigator — National University of Ireland, Galway
Locations (1):
- Physiology laboratory, Galway, Galway, Ireland

REFERENCES:
- [Background] Rating D, Langhans CD. Breath tests: concepts, applications and limitations. Eur J Pediatr. 1997 Aug;156 Suppl 1:S18-23. doi: 10.1007/pl00014264. PMID 9266210
- [Background] Stellaard F, Koetse HA, Elzinga H, Boverhof R, Tjoonk R, Klimp A, Vegter D, Liesker J, Vonk RJ. 13C-carbohydrate breath tests: impact of physical activity on the rate-limiting step in lactose utilization. Scand J Gastroenterol. 2000 Aug;35(8):819-23. doi: 10.1080/003655200750023183. PMID 10994620
- [Background] Lifschitz CH, Boutton TW, Carrazza F, Beyreiss K, Schmitz J, Ricour C, Shulman R, Nichols BL. A carbon-13 breath test to characterize glucose absorption and utilization in children. J Pediatr Gastroenterol Nutr. 1988 Nov-Dec;7(6):842-7. doi: 10.1097/00005176-198811000-00008. PMID 3143819
- [Background] Mizrahi M, Lalazar G, Adar T, Raz I, Ilan Y. Assessment of insulin resistance by a 13C glucose breath test: a new tool for early diagnosis and follow-up of high-risk patients. Nutr J. 2010 May 27;9:25. doi: 10.1186/1475-2891-9-25. PMID 20507559
- [Background] Dillon EL, Janghorbani M, Angel JA, Casperson SL, Grady JJ, Urban RJ, Volpi E, Sheffield-Moore M. Novel noninvasive breath test method for screening individuals at risk for diabetes. Diabetes Care. 2009 Mar;32(3):430-5. doi: 10.2337/dc08-1578. Epub 2008 Dec 15. PMID 19074994